CLINICAL TRIAL: NCT05997173
Title: The Regulatory Role of Immune Response in Oral Lichen Planus With Mental Disorders
Brief Title: The Regulatory Role of Immune Response in Oral Lichen Planus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BMU81800920402
Record Dates: First submitted 2023-07-15; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-09

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; depression; anxiety; mesenchymal stem cells
MeSH Terms: conditions — Lichen Planus, Oral; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Normal control group
  Interventions: Other: Control
- Non erosive OLP: Non erosive oral lichen planus
  Interventions: Other: Non erosive OLP
- Erosive OLP: Erosive oral lichen planus
  Interventions: Other: Erosive OLP

INTERVENTIONS:
Other: Control — Investigation of scale of control
  Groups: Control
Other: Non erosive OLP — Investigation of cale of non erosive OLP patients
  Groups: Non erosive OLP
Other: Erosive OLP — Investigation of cale of erosive OLP patients
  Groups: Erosive OLP

SUMMARY:
Oral lichen planus (OLP) is a common chronic inflammatory disease of Oral mucosa. The pathogenesis of OLP is not clear, and there is no effective method to cure it. In vitro, previous studies have shown that oral mucosal mesenchymal stem cell cells (MSCs) can secrete Ido, which is involved in the pathogenesis of OLP. It has been proved that mental disorders such as depression and anxiety play an important role in the pathogenesis and treatment of OLP. Mental stress factors can cause abnormal changes of inflammatory factors, leading to immune dysfunction, which is also one of the main causes of OLP. In this study, we integrated the advantages of stomatology, psychiatry, neurobiology and traditional Chinese medicine, focused on the clinical problems of mental disorders with oral mucosal comorbidity, and assessed the depressive and anxiety status of OLP patients, so as to improve the therapeutic effect of OLP.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral lichen planus
* male or female patients older than 18 years of age
* patients willing to participate with signed informed consent.

Exclusion Criteria:

* pregnant or lactating
* had serious systemic diseases of the heart, lung, liver, and kidney, or had tumors
* were unwilling to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with oral lichen planus or control Male or female patients older than 18 years of age Participants willing to participate with signed informed consent.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The scores of the scale with the symptoms and signs of the disease | During the initial diagnosis，through study completion, an average of 1 year
  Psychological factors in OLP patients and normal controls were assessed using psychological scales such as the Hamilton Anxiety Scale (HAMA) and Hamilton Depression Scale (HAMD). Tissue and blood samples were collected during visits, and the concentrations of inflammatory factors in normal and lesion tissues were detected using immunofluorescence, flow cytometry, and enzyme-linked immunosorbent assay (ELISA). Statistical analysis was performed to determine the correlation between emotional disorders and inflammation in OLP patients, aiming to elucidate the underlying pathogenic mechanisms.

SECONDARY OUTCOMES:
Immune inflammatory response | During the initial diagnosis，through study completion, an average of 1 year
  Psychological factors in OLP patients and normal controls were assessed using psychological scales such as the Hamilton Anxiety Scale (HAMA) and Hamilton Depression Scale (HAMD). Tissue and blood samples were collected during visits, and the concentrations of inflammatory factors in normal and lesion tissues were detected using immunofluorescence, flow cytometry, and enzyme-linked immunosorbent assay (ELISA). Statistical analysis was performed to determine the correlation between emotional disorders and inflammation in OLP patients, aiming to elucidate the underlying pathogenic mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihui Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashmi AM, Butt Z, Umair M. Is depression an inflammatory condition? A review of available evidence. J Pak Med Assoc. 2013 Jul;63(7):899-906. PMID 23901717
- [Background] Alrashdan MS, Cirillo N, McCullough M. Oral lichen planus: a literature review and update. Arch Dermatol Res. 2016 Oct;308(8):539-51. doi: 10.1007/s00403-016-1667-2. Epub 2016 Jun 27. PMID 27349424
- [Background] Thapar A, Collishaw S, Pine DS, Thapar AK. Depression in adolescence. Lancet. 2012 Mar 17;379(9820):1056-67. doi: 10.1016/S0140-6736(11)60871-4. Epub 2012 Feb 2. PMID 22305766
- [Background] Nitzan U, Carmeli G, Chalamish Y, Braw Y, Kirsch I, Shefet D, Krieger I, Mendlovic S, Bloch Y, Lichtenberg P. Open-Label placebo for the treatment of unipolar depression: Results from a randomized controlled trial. J Affect Disord. 2020 Nov 1;276:707-710. doi: 10.1016/j.jad.2020.07.077. Epub 2020 Jul 21. PMID 32871704
- [Background] Vilar-Villanueva M, Gandara-Vila P, Blanco-Aguilera E, Otero-Rey EM, Rodriguez-Lado L, Garcia-Garcia A, Blanco-Carrion A. Psychological disorders and quality of life in oral lichen planus patients and a control group. Oral Dis. 2019 Sep;25(6):1645-1651. doi: 10.1111/odi.13106. Epub 2019 May 29. PMID 30993798